CLINICAL TRIAL: NCT03054675
Title: Perioperative Lung Function Monitoring After Anatomic Lung Resections
Acronym: PLF
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 266/15
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Lung Function Decreased; Lung Diseases; Surgery
Keywords: lung resection; lung function; VATS; Thoracotomy
MeSH Terms: conditions — Respiratory Insufficiency; Lung Diseases | interventions — Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pneumonia: Patients suffering from postoperative pneumonia including all three of the following:
  1. Clinical signs of a pulmonary infection (i.e. fever ≥ 38°C combined with productive cough and/or dyspnea)
  2. A new rise of inflammatory markers (i.e. WBC count ≥ 10.5 x 109 and elevated CRP)
  3. New radiographic infiltrates on chest x-ray without another explanation. Patients with pneumonia undergo spirometry before and on every second day after lung surgery
  Interventions: Diagnostic Test: Spirometry
- No Pneumonia: Patients without pneumonia undergo spirometry before and on every second day after lung surgery
  Interventions: Diagnostic Test: Spirometry
- Open (no pneumonia): Patients undergoing open anatomical lung resection who did not show postoperative pneumonia.
  All patients undergo spirometry before and on every second day after lung surgery.
  Interventions: Diagnostic Test: Spirometry
- Minimally invasive (no pneumonia): Patients undergoing minimally invasive anatomical lung resection who did not show postoperative pneumonia.
  All patients undergo spirometry before and on every second day after lung surgery.
  Interventions: Diagnostic Test: Spirometry

INTERVENTIONS:
Diagnostic Test: Spirometry — Absolute FEV1 is measured in every patient using a handheld spirometer

SUMMARY:
Aim of this study was to prospectively investigate the correlation between postoperative spirometry values and pulmonary complications after anatomic lung resections. In addition, the investigators compared postoperative pulmonary function changes between open and minimally invasive approaches.

DETAILED DESCRIPTION:
All patients undergoing an anatomical lung resection at the investigators' institution were evaluated for this study. Underage patients and those undergoing extended resections (including resection of the chest wall and/or diaphragm) and/or bronchoplastic procedures were excluded.

In every eligible patient undergoing an anatomic lung resection, preoperative spirometry was performed using a handheld spirometer on the day before surgery and on every second day after surgery was performed until patient discharge. The absolute values of FEV1 were recorded by an independent study nurse and noted on a separate sheet not available to the treating doctors.

At the end of the study period FEV1 values were evaluated especially with focus on their correlation with postoperative pulmonary complications (i.e. pneumonia, acute exacerbation of COPD, air leak and atelectasis). Furthermore lung function values of patients undergoing 'open' resections were compared with patients undergoing minimally invasive resections.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing anatomical lung resection
* Written informed consent

Exclusion Criteria:

* Underage patients
* Extended resections including resection of chest wall or diaphragm
* Bronchoplastic resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing an anatomical lung resection at our institution
Sampling Method: Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Decrease in FEV1 | up to 6 days after surgery
  Postoperative loss of FEV1 in percent of absolute preoperative levels

CONTACTS AND LOCATIONS:
Overall Officials: Gregor J Kocher, MD, Principal Investigator — Division of General Thoracic Surgery, University Hospital Bern
Locations (1):
- University Hospital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ercegovac M, Subotic D, Zugic V, Jakovic R, Moskovljevic D, Bascarevic S, Mujovic N. Postoperative complications do not influence the pattern of early lung function recovery after lung resection for lung cancer in patients at risk. J Cardiothorac Surg. 2014 May 19;9:92. doi: 10.1186/1749-8090-9-92. PMID 24884793
- [Background] Nakata M, Saeki H, Yokoyama N, Kurita A, Takiyama W, Takashima S. Pulmonary function after lobectomy: video-assisted thoracic surgery versus thoracotomy. Ann Thorac Surg. 2000 Sep;70(3):938-41. doi: 10.1016/s0003-4975(00)01513-7. PMID 11016337
- [Result] Schussler O, Alifano M, Dermine H, Strano S, Casetta A, Sepulveda S, Chafik A, Coignard S, Rabbat A, Regnard JF. Postoperative pneumonia after major lung resection. Am J Respir Crit Care Med. 2006 May 15;173(10):1161-9. doi: 10.1164/rccm.200510-1556OC. Epub 2006 Feb 10. PMID 16474029